CLINICAL TRIAL: NCT07078708
Title: Effectiveness of Non-hormonal Treatment on Moderate to Severe Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haleema Sadia (Other)
Responsible Party: Sponsor-Investigator, Haleema Sadia, Dr Haleema Sadia, Avicenna Medical College Lahore
Organization: Avicenna Medical College Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Premenstrual Syndrome-PMS
Keywords: Calcium; Vitamin-D; Premenstrual Symptoms
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Vitamin D; Cholecalciferol; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants taking calcium and Vitamin D (Experimental): In this group participants received vitamin D supplementation at a dose of 50,000 IU every two weeks along with a daily intake of 1,000 mg of calcium for 12 weeks. Participants symptoms were assessed at baseline, one month, three months, and six months following the commencement of the study.
  Interventions: Dietary Supplement: vitamin D (cholecalciferol) supplementation
- Participants taking placebo (Placebo Comparator): In this group participants received placebo for 12 weeks. Participants symptoms were assessed at baseline, one month, three months, and six months following the commencement of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D (cholecalciferol) supplementation — Vitamin D supplementation at a dose of 50,000 IU every two weeks along with a daily intake of 1,000 mg of calcium for 12 weeks
  Arms: Participants taking calcium and Vitamin D
Other: Placebo — Placebo was given for 12 weeks
  Arms: Participants taking placebo

SUMMARY:
A double-blind, randomised, placebo-controlled, parallel trial was conducted involving 100 females aged 18-40, all of whom presented with premenstrual syndrome at the Department of Gynecology and Obstetrics, Avicenna Medical College Hospital, Lahore, Pakistan. Participants were randomly assigned to two groups of equal size: One group received vitamin D supplementation at a dose of 50,000 IU every two weeks along with a daily intake of 1,000 mg of calcium, whereas the comparison group was administered a placebo under the same conditions for 12 weeks. All the participants were examined on premenstrual syndrome with the Premenstrual Symptoms Screening Tool-Adolescent (PSST-A) questionnaire

DETAILED DESCRIPTION:
A double-blind, randomised, placebo-controlled, parallel trial was conducted involving 100 females aged 18-40, all of whom presented with premenstrual syndrome at the Department of Gynecology and Obstetrics, Avicenna Medical College Hospital, Lahore, Pakistan. Participants were randomly assigned to two groups of equal size: One group received vitamin D supplementation at a dose of 50,000 IU every two weeks along with a daily intake of 1,000 mg of calcium, whereas the comparison group was administered a placebo under the same conditions for 12 weeks. All the participants were examined on premenstrual syndrome with the Premenstrual Symptoms Screening Tool-Adolescent (PSST-A) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-40 years with moderate to severe PMS

Exclusion Criteria:

* Individuals exhibiting symptoms of malnutrition or requiring calcium+vitamin D supplementation.
* Individuals with systemic diseases such as sepsis, hemodynamic instability, or acute meningitis; diarrhoea.
* Individuals with known intolerance or sensitivity to calcium vitamin D or calcium vitamin D containing compounds.
* smokers, Individuals with exposure to stressful situations or a history of mental illness.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Depressed mood | 6 Months
  Outcome was assessed by using Premenstrual Symptoms Screening Tool-Adolescent (PSST-A) questionnaire in both groups and analyzed.

SECONDARY OUTCOMES:
Decreased interest in work activities | 6 Months
  Outcome was assessed by using Premenstrual Symptoms Screening Tool-Adolescent (PSST-A) questionnaire in both groups and analyzed.
Difficulty in concentration | 6 Months
  Outcome was assessed by using Premenstrual Symptoms Screening Tool-Adolescent (PSST-A) questionnaire in both groups and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenna Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No